CLINICAL TRIAL: NCT05894811
Title: A Study on the Effect of Bariatric Surgery on Glucose Metabolism in Chinese Obese and Type 2 Diabetes Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Dongyang Liu (Other)
Responsible Party: Sponsor-Investigator, Dongyang Liu, researcher, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: DCTC-IIR202307
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Diabete Type 2; Obesity
Keywords: Diabete Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: obese people with normal glucose tolerance
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI
- IGT: obese people with injured glucose tolerance
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI
- T2D: obese people with type 2 diabetes
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — Nine blood samples were collected from subjects within 4 hours of oral glucose administration, 0 min before oral glucose administration, and 10, 20, 30, 60, 90, 120, 180, 240 min afterwards, and 4 mL of venous blood was collected at each time point for glucose, C-peptide and insulin concentrations.
Diagnostic Test: MRI — Using MRI to quantify of fat content in the liver and pancreas of the subjects

SUMMARY:
The study will be conducted in the following population: obese patients with normal glucose tolerance (HbA1c ≤ 5.6%, n=12), pre-sugar patients (5.7% ≤ HbA1c ≤ 6.4%, n=18) and patients with T2DM (HbA1c ≥ 6.4% , n=18). After recruiting, they were followed up at 1, 3, 6, and 12 months postoperatively, and their preoperative and follow-up examination values related to demographics, body composition, blood biochemistry, and glucose metabolic balance, as well as quantitative MRI imaging and oral glucose tolerance test (OGTT) will be collected. An interim analysis will be performed at 6 months postoperatively and overall analysis will be performed at 12 months postoperatively by descriptive statistics and ANOVA methods to explore the effect of adiposity on the progression of diabetes mellitus and insulin secretory function.

DETAILED DESCRIPTION:
The study will be conducted in the following population: obese patients with normal glucose tolerance (HbA1c ≤ 5.6%, n=12), pre-sugar patients (5.7% ≤ HbA1c ≤ 6.4%, n=18) and patients with T2DM (HbA1c ≥ 6.4% , n=18). After recruiting, they were followed up at 1, 3, 6, and 12 months postoperatively, and their preoperative and follow-up examination values related to demographics, body composition, blood biochemistry, and glucose metabolic balance, as well as quantitative MRI imaging and oral glucose tolerance test (OGTT) will be collected. An interim analysis will be performed at 6 months postoperatively and overall analysis will be performed at 12 months postoperatively by descriptive statistics and ANOVA methods to explore the effect of adiposity on the progression of diabetes mellitus and insulin secretory function.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 28 kg/m2, meeting the indications for surgical weight loss surgery (gastrectomy)
* Normal glucose tolerance group: HbA1c ≤ 5.6%; ≥ 6 cases aged 24 years or above
* IGT patients: 5.7% ≤ HbA1c ≤ 6.4%; ≥ 12 cases aged 24 years or above
* T2DM patients: Subjects with HbA1c ≥ 6.4% or HbA1c well controlled by medication can be diagnosed as T2DM based on self-reported or fasting/postprandial blood glucose diagnosis; ≥ 12 cases aged 24 years and above.
* Between the ages of 16 and 65 (inclusive), with no less than one-third of either gender
* The subjects understand the content of the informed consent form and voluntarily sign it, which allows them to maintain good communication with the researchers and comply with the requirements of the clinical trial

Exclusion Criteria:

* Type I diabetes patients (autoimmune diabetes patients with T1DM antibody)
* Suffering from special types of diabetes, including cortisolism, growth hormone tumor, glucagon tumor and diabetes caused by some genetic factors
* Significant weight loss occurred before enrollment (>3% weight loss in the first 3 months)
* Participated in other research projects as a subject within 6 months prior to screening
* Donate or lose ≥ 400 mL of blood within 8 weeks prior to screening
* Regular use (cumulative use for 3 months in the past 12 months) or treatment with corticosteroids, contraceptives, thiazide diuretics, and quinolone antibiotics in the past two months
* Regular use (cumulative use for 3 months in the past 12 months) or treatment with anti obesity drugs in the past two months
* The following hypoglycemic drugs have been used routinely (for 3 months accumulatively in the past 12 months) or in the past two months: sulfonylureas (glibenclamide, glipizide, gliclazide, gliquidone, glimepiride, etc.), non sulfonylureas (repaglinide, nateglinide, migglinide, etc.), GLP-1 receptor agonists (exenatide, lilalutide, etc.) DPP-4 inhibitors (sigliptin, alogliptin, vildagliptin, shagliptin, linagliptin, etc.) or glucokinase agonists (doegliptin, etc.)
* Contraindications to magnetic resonance imaging
* The risk of complications significantly increases during the perioperative or postoperative period
* Those with a history of other weight loss surgeries
* Individuals with a history of cardiovascular surgery and severe cardiovascular and pulmonary diseases: including stroke, severe coronary heart disease, arrhythmia, unstable angina, myocardial infarction within 6 months, peripheral vascular disease, heart failure, and uncontrolled hypertension
* Clinically significant history of ECG abnormalities or family history of long QT syndrome (grandparents, parents, brothers and sisters)
* People with a history of kidney disease: have a history or evidence of renal insufficiency, manifested as clinically significant creatinine abnormalities or urinary composition abnormalities (such as tubular abnormalities), or eGFR<60 ml/min/1.73m2
* Patients with a history of gastrointestinal surgery (excluding appendectomy and cholecystectomy), inflammatory bowel disease, esophageal disease, including severe refractory esophagitis, Barrett's disease, esophageal motility disorders, or other gastric motility impairments, or those with esophageal hiatal hernia>3cm in size, chronic or acute bleeding, including peptic ulcer disease, portal hypertension (gastric or esophageal varices), chronic pancreatitis or cirrhosis
* Individuals with a history of eating disorders or mental illness
* Individuals with a history of infectious diseases are excluded if they have any of the following: human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or those who have tested positive for syphilis
* Smokers, those who smoke more than 10 cigarettes or equivalent amounts of tobacco per day and cannot stop smoking during the trial period
* There is a history of drug or alcohol abuse within the 12 months prior to the trial, or evidence of such abuse is found during laboratory examinations during the screening period evaluation
* Women who are pregnant, breastfeeding, or planning to conceive and are unwilling to use contraception during the trial period
* Malignant tumor patients
* The researcher believes that it is not suitable for participants in the experiment
* For different types of subjects, additional exclusion criteria: obese patients with normal glucose tolerance: fasting blood glucose ≥ 7.0 mmol/L or ≤ 3.9 mmol/L (excluding diabetes and hypoglycemia)
* Obese patients before glucose: fasting blood glucose ≥ 7.0 mmol/L or ≤ 3.9 mmol/L (excluding diabetes and hypoglycemia)
* Obese T2DM patients: Fasting blood glucose ≤ 3.9 mmol/L (excluding those with hypoglycemia)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese people who will undergo sleeve gastrectomy in Peking University Third Hospital and meet the admission criteria.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Visceral fat content | 1 day
  Visceral fat content (MRI)
Islet function indicators | 1 day
  indicators describing Islet function calculated from OGTT data using MTT model

IPD SHARING:
Plan to Share IPD: No